CLINICAL TRIAL: NCT02103738
Title: Canadian Treat and Extend Analysis Trial With Ranibizumab
Acronym: CAN-TREAT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002ACA06
Record Dates: First submitted 2014-02-18; First posted 2014-04-04 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: wetAMD
Keywords: Lucentis; Ranibizumab; Treat and Extend; wetAMD; Age related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1 (Monthly): 0.5 mg intravitreal injections of Ranibizumab monthly for the duration of the study.
  Interventions: Other: 0.5 mg Ranibizumab intravitreal injections
- Arm 2 (Treat and Extend): Three consecutive months of 0.5 mg Ranibizumab intravitreal injections (Day 1, Month 1, and Month 2). Monthly injections will continue until evidence of disease stability is observed. Specifically, monthly treatment will continue until visual acuity is deemed stable as indicated by a gain in visual acuity of ≤ 3 ETDRS letters from the prior month, no clinical evidence of lesion growth, fluid or blood, and no intraretinal or subretinal fluid on OCT. When this is achieved, the intervals between each subsequent injection will be extended by 2 weeks (intervals of 6 weeks, 8 weeks, 10 weeks, to a maximum of 12 weeks) until clinical or diagnostic evidence of disease instability is observed based on OCT findings and/or BCVA ETDRS.
  Interventions: Other: 0.5 mg Ranibizumab intravitreal injections

INTERVENTIONS:
Other: 0.5 mg Ranibizumab intravitreal injections — All eligible patients will initially be treated in a fixed loading phase, consisting of one intravitreal injection of Ranibizumab 0.5 mg per month for 3 consecutive months (Day 1, Month 1, and Month 2). After the loading phase, patients will be treated according to the treatment arm to which they have been assigned, either a continued once monthly dosing regimen, or an extended schedule of Ranibizumab intravitreal injections as described below. The planned duration of total treatment is 24 months.

SUMMARY:
This is an observational study to will evaluate and compare two Ranibizumab treatment regimens (Standard of care) in patients with neovascular (wet) age-related macular degeneration (wAMD) aiming to achieve and to maintain a maximum visual function benefit. The results will be used to generate further recommendations on the timing of treatment administration for patients with neovascular (wet) age-related macular degeneration (wAMD). In this context, the study will use the anatomical imaging (for example, optical coherence tomography [OCT]) to evaluate wAMD disease activity impacted by the recurrence of disease instability and for decision making in the treatment decision algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Infomed consent,
* Male and Female, 50 years of age or older
* Diagnosis of treatment-naive CNV secondary to age-related macular degeneration(AMD) in the study eye,
* BCVA score between 78 and 19 letters inclusive,

Exclusion Criteria:

* Patients with structural foveal damage in the study eye,
* Patients with confounding severe oculare diseases,
* Patients with suspicion of ( Polypoidal Choroidal Vasculapathy PCV) in the study eye,
* Patients with active or suspected or periocular infections in either eye or active intraocular inflammation in either eye,
* Patients who had previous subfoveal laser photocoagulation in the study eye or history of vitrectomy surgery in the study eye,
* Patients who had any prior treatment in the study eye, e.g., with Visudyne*, Avastin*, prior Ranibizumab treatment, Ozurdex*, external radiation therapy, transpupillary thermotherapy (TTT), or any intravitreal injection,
* Patients with a known sensitivity to Ranibizumab or any component of its formulation,
* Patients who have used any investigational agent in the last 30 days,
* Concurrent participation in a clinical trial or within 30 days prior to enrollment,
* Patients having received systemic treatment with any other anti-vascular endothelial growth factor (VEGF) therapy ≤ 60 days prior to enrollment
* Patients with physical or mental disabilities that prevent accurate vision testing,
* Patients physically unable to tolerate intravenous fluorescein angiography,
* Pregnant or breastfeeding female patients,
* Any patient with recent history of new onset cardiac disease or thromboembolic central nervous system (CNS) event (within 12 months of Baseline Visit),
* Patients with any other condition which, in the opinion of the Investigator, would require treatment that would significantly impact the treatment assessments during this study.

Ages: 50 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of male and female Canadian patients diagnosed with visual impairment due to wAMD and for whom Ranibizumab has been prescribed as their standard of care by the treating physician. Eligibility for Ranibizumab will be determined by the study physician according to the current prescribing information. A total of 580 patients will be enrolled from approximately 20 to 25 centers.
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Mean Change in Visual Acuity | Baseline to Month 12
  Visual Acuity (VA) will be assessed using best correction determined from protocol refraction during screening and every 3 months throughout the study; in the monthly regimen and during screening and at every visit thereafter throughout the study in the treat and extend regimen. VA measurements (number of letters correctly identified) will be performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like VA testing charts at an initial testing distance of 4 meters. This outcome measure will describe the difference in the VA mean changes between the two regimens from Baseline to Month 12.

SECONDARY OUTCOMES:
Proportion of patients with a gain of equal or more than 5, 10, and 15 letters between the 2 treatment arms. | Baseline to Month 12
Proportion of patients with a gain of equal or more than 5, 10, and 15 letters between the 2 treatment arms. | Baseline to Month 24
Proportion of patients with a loss of less than 5, 10, and 15 letters between the 2 treatment arms from baseline to Month 12 and from baseline to Month 24. | baseline to Month 12
Proportion of patients with a loss of less than 5, 10, and 15 letters between the 2 treatment arms. | baseline to Month 24
Mean change in BCVA ETDRS between the 2 treatment arms at Month 12 compared to Month 3. | Month 12 and Month 3
Mean change in BCVA ETDRS between the 2 treatment arms. | Baseline to Month 24
Number of injections performed in each treatment arms. | Baseline to Month 24
Number of injections performed in each treatment arms. | Month 12 to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Canada (17):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Missisauga, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Timmins, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Drummondville, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Thetford-Mines, Quebec

REFERENCES:
- [Derived] Kertes PJ, Galic IJ, Greve M, Williams G, Baker J, Lahaie M, Sheidow T. Efficacy of a Treat-and-Extend Regimen With Ranibizumab in Patients With Neovascular Age-Related Macular Disease: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 Mar 1;138(3):244-250. doi: 10.1001/jamaophthalmol.2019.5540. PMID 31917441